CLINICAL TRIAL: NCT05947955
Title: A Phase 2 Randomized Double-blind Placebo-controlled Study To Evaluate The Efficacy And Safety Of Adjunctive Recombinant Human Plasma Gelsolin With Standard Care For Moderate-to-Severe ARDS Due To Pneumonia Or Other Infections
Brief Title: Rhu-pGSN for Acute Respiratory Distress Syndrome (ARDS)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioAegis Therapeutics Inc. (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTI-203
Record Dates: First submitted 2023-07-09; First posted 2023-07-17 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Acute Respiratory Distress Syndrome; Infections
Keywords: moderate to severe ARDS; respiratory failure; rhu-pGSN
MeSH Terms: conditions — Respiratory Distress Syndrome; Infections; Respiratory Insufficiency | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: 1:1 randomization to rhu-pGSN or saline placebo arm
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The placebo of normal saline is visibly indistinguishable from the study drug ans is to be at the same volume of administration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rhu-pGSN Treatment (Experimental): Subjects will receive rhu-pGSN 24 mg/kg once, followed by 5 daily doses of 12 mg/kg based on actual body weight in addition to standard care .
  Interventions: Drug: Rhu-pGSN
- Normal Saline Placebo (Placebo Comparator): Subjects will receive 6 doses of normal-saline placebo in volumes equivalent to subjects given rhu-pGSN in addition to standard care.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Rhu-pGSN — Intravenous administration based on actual body weight
  Other Names: recombinant human gelsolin
  Arms: Rhu-pGSN Treatment
Drug: normal saline — intravenous administration in the same volume as the active therapy
  Other Names: 0.9% sterile saline
  Arms: Normal Saline Placebo

SUMMARY:
BTI-203 is a randomized, double-blind, placebo-controlled, multicenter, Phase 2 proof-of-concept (POC) study to evaluate the efficacy and safety of rhu-pGSN plus standard of care (SOC) in subjects with moderate-to-severe ARDS (P/F ratio ≤150) due to pneumonia or other infections. Potential subjects hospitalized with pneumonia or other infections are to be screened within 24 hours of diagnosis of ARDS.

DETAILED DESCRIPTION:
Potential subjects hospitalized with pneumonia or other infections are to be screened within 24 hours of diagnosis of ARDS. The Sponsor aims to identify as early as possible patients in the hospital who have developed acute hypoxemic respiratory failure within 7 days of the precipitating infection (often fever, rigors, chills, increased heart rate, increased respiratory rate, pain, cough, etc.) leading to ARDS resulting in mechanical or noninvasive ventilation or high-flow nasal oxygen (HFNO) supplementation with ≥50% O2 at a flow rate of ≥30 L/min. Patients who do not qualify for the study at the initial screening visit because of mild ARDS may subsequently progress to moderate-to-severe ARDS and should be reassessed at least daily for the 7 days following the precipitating infection.

Once informed consent is obtained, the following assessments/procedures will be performed:

1. Confirm the potential participant has acute hypoxemic respiratory failure qualifying as moderate-to-severe ARDS for ≤48 hours following a suspected or confirmed infection within the preceding week. Moderate-to-severe ARDS is defined by the calculated or estimated ratio of arterial pressure of O2 to the fraction of inspired O2 [P/F ratio] ≤150. The P/F ratio will be computed from the most recent arterial blood gas obtained no more than 12 hours earlier than randomization. For potential subjects on high-flow nasal oxygen with ≥50% O2 at a flow rate of ≥30 L/min, the P/F ratio will be estimated assuming 50% delivered O2. If eligible and entered in the trial, the following steps should be taken.
2. Record medical history, including concomitant medications and current clinical status. Specify the site and etiology (if known) of infection, indicating if the lung ("direct ARDS") or another organ ("indirect ARDS") is the primary site of infection.
3. Perform pregnancy test (urine or blood) for women of childbearing potential if not already performed during the current hospitalization.
4. Collect pretreatment blood samples for measurement of baseline pGSN and analysis of antibodies against pGSN.
5. Perform physical examination and document results of the chest x-ray (CXR) and/or computed tomography (CT) scan, if CXR is inadequate if not already available as per SOC.
6. Obtain blood and sputum cultures and electrocardiogram (EKG) per SOC (if not already performed). Document the site of infection by collecting specimens as indicated: sputum (bacterial, viral, and mycobacterial, as indicated) and blood cultures, sputum Gram-stains, antigen detection on respiratory and urine specimens, and syndromic nucleic acid amplification tests (NAATs) on respiratory specimens (including a viral and other respiratory pathogen polymerase chain reaction [PCR] panel), where possible. Other specimens from possible sites of infection (e.g., urine, intra-abdominal drainage, skin or soft-tissue abscesses) should be cultured when available.
7. Measure routine lab tests at local (hospital) laboratory per local custom/SOC collect aliquots f- blood for subsequent biomarker assays (including, but not limited to C-reactive protein [CRP], procalcitonin, interleukin [IL]1β, IL6, IL10, and tumor necrosis factor [TNF]) for analysis at the central laboratory.
8. If eligibility criteria are satisfied, the subject will be randomized 1:1 (rhu-pGSN:placebo) by site to a treatment group and treated within 12 hours of randomization and no later than 48 hours after the diagnosis of moderate-to-severe ARDS.

Randomized subjects will receive the assigned dose of rhu-pGSN or an equal volume of visibly indistinguishable sterile saline placebo as soon as possible but beginning no later than 48 hours after the diagnosis of moderate-to-severe ARDS. After reconstitution, rhu-pGSN is not to be kept at room temperature for >2 hours prior to beginning study drug administration.

A single loading dose of rhu-pGSN at 24 mg/kg followed by 5 daily doses of rhu-pGSN at 12 mg/kg of measured or estimated actual body weight starting 24 hours after the loading dose or an equal volume of indistinguishable saline placebo will be administered. A window of ±2 hours will be allowed around dosing times. Study drug is administered by an IV push through a 0.2 μm filter. The syringe, filter, and extension tubing for administration of study drug are to be connected as close to the subjects as possible.

The primary efficacy endpoint of all-cause mortality will be assessed at Day 28. All-cause mortality will also be assessed on Days 7 and 14. Discharged subjects will undergo follow-up evaluation on Days 14 and 28, preferably but not necessarily in person. Survival at Day 60 will be confirmed by telephonic contact or after 3 failed attempts, review of hospital and public records that document survival or death.

Screening laboratory and other tests may be used as baseline values and do not need to be repeated if performed within 24 hours prior to randomization unless otherwise dictated by SOC. However, the blood sample for analysis of pGSN levels is to be repeated if not collected within 15 minutes before initiating the first dose of study drug.

Repeat CXRs and/or CT scans and labs/cultures are to be obtained during the hospitalization if/when indicated by SOC. On Days 1 (predose) and 28, blood samples for analysis of antibodies against pGSN are to be collected, if possible. Repeat blood and other cultures should be obtained per SOC.

An independent Data and Safety Monitoring Board (DSMB) consisting of at least 2 physicians and 1 statistician with appropriate scientific and medical expertise will be formed, and its roles and responsibilities will be described in the DSMB charter. The DSMB will perform 5 periodic reviews of safety data emphasizing deaths and SAEs and will monitor stopping rules to pause enrollment. There will be no pause on enrollment during the planned unblinded periodic reviews. These reviews will be performed after the first 50, 100, 200, 300, and 400 subjects in the Safety Analysis Set have either completed 28 days of follow-up, have died, or have discontinued from the study prior to completing 28 days of follow-up. DSMB members will be provided with unblinded data. Based on the results of each of the planned periodic reviews, the study will be paused only if there is a relative increase of 25 percentage points in the incidence of death or SAEs in the rhu-pGSN treatment group compared to the placebo group. A futility analysis will be performed at the 300-subject review. The Sponsor will take appropriate action based on the recommendation of the DSMB.

The DSMB will also review expedited reports of any SAEs throughout the study and may request additional looks at safety data at their discretion. Enrollment will continue during all safety analyses unless otherwise recommended by the DSMB chair.

ELIGIBILITY:
Inclusion Criteria:

1. Infection followed within a week of documented bilateral infiltrates/opacities consistent with ARDS, as assessed by the admitting emergency department, clinic, intensivist, or ward physician or equivalent caregiver or a radiologist

   * Investigator or designee to note radiologic findings in the electronic case report form (eCRF)
   * Radiology report and conclusion should be summarized in the eCRF
   * A digital copy of the radiograph uploaded and saved for review
2. Acute hypoxemic respiratory failure (moderate-to-severe ARDS) for ≤48 hours associated with suspected or confirmed infection (moderate-to-severe ARDS defined by the ratio of arterial pressure of O2 to the fraction of inspired O2 ≤150). Eligible subjects will be intubated for mechanical ventilation, receiving noninvasive ventilation by continuous positive airway pressure (CPAP) or bilevel positive airway pressure (BiPAP), or on HFNO at least 30 L/min of 50% or greater inspired O2. Although it is expected that most eligible subjects will be receiving positive end-expiratory pressure (PEEP) or CPAP ≥5 cm H2O consistent with the original Berlin definition (ARDS Definition Task Force 2012), these measures will not be mandated as entry criteria.
3. Age ≥18 years
4. Informed consent obtained from subject/next of kin/legal proxy
5. Clear or convincing evidence of a precipitating infection during the 7 days preceding the diagnosis of ARDS in the judgement of the screening or primary care team
6. During the course of the study starting at screening and for at least 3 months after their final study treatment:

   1. Female subjects of childbearing potential must agree to use 2 medically accepted and approved birth control methods
   2. Male subjects with a partner who might become pregnant must agree to use reliable forms of contraception (i.e., vasectomy, abstinence), or an acceptable method of birth control must be used by the partner
   3. All subjects must agree not to donate sperm or eggs

Exclusion Criteria:

1. Ongoing evidence or suspicion that heart failure, volume overload, pulmonary emboli, atelectasis, chronic lung disease, pleural effusion, cardiac tamponade, or constrictive pericarditis are materially contributing to the clinical or radiological findings bas assessed by the care team or Investigator; an echocardiogram is strongly recommended as part of standard care to exclude a significant contribution of systolic or diastolic heart failure and volume overload.
2. Presence of systemic fungal, yeast, parasitic, or mycobacterial infection
3. Current or planned receipt of extracorporeal membrane oxygenation (ECMO)
4. Pregnant or lactating women
5. Previous splenectomy
6. Any vaccination in the previous 30 days
7. Participation in an investigational clinical trial (e.g., device, drug, or biologic) in the previous 30 days
8. Known allergy to study drug or excipients
9. Weight >125 kg
10. Active underlying cancer or treatment with systemic chemotherapy or radiation therapy during the last 60 days or likely to require similar treatments during the ensuing 6 months
11. Transplantation of hematopoietic or solid organs, graft versus host disease, or post-transplant lymphoproliferative disease
12. Chronic mechanical ventilation or dialysis
13. Unsuitable for study participation, in the opinion of the Investigator, because of chronic, severe, end-stage, or life-limiting underlying disease unrelated to current infection likely to interfere with management and assessment of ARDS, only comfort or limited (non-aggressive) care is to be given, or life expectancy <6 months unrelated to acute infection in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality at day 28 | 28 days
  Death for any reason through Day 28 between treatment groups

SECONDARY OUTCOMES:
Ventilator-free days | 28 days
  Ventilator-free days through Day 28 between treatment groups
All-cause mortality at day 60 | 60 days
  Death for any reason through Day 60 between treatment groups
Proportion of surviving subjects without respiratory support | 28 days
  Proportion of surviving subjects without respiratory support over time (Days 7, 14, and 28) between treatment groups
Time to death and proportions of subjects dying over time | 28 days
  Time to death and proportions of subjects dying over time (Days 7, 14, and 28) between treatment groups
Time to discontinuation of respiratory support and proportions without respiratory support | 28 days
  Time to discontinuation of respiratory support and proportions without respiratory support over time (Days 7, 14, and 28) between treatment groups
Frequency of intubation | 28 days
  For subjects not intubated at entry, the frequency of intubation through Day 28 between treatment groups
Days in the ICU and in the hospital | 28 days
  Days in the ICU and in the hospital through Day 28 between treatment groups
Frequency of RRT | 28 days
  Frequency of renal replacement therapy (RRT) through Day 28 between treatment groups
SAEs and AEs | 28 days
  Incidence, causality, and severity of SAEs and AEs (graded according to the NCI CTCAE version 5.0 [or higher]) between treatment groups

CONTACTS AND LOCATIONS:
Locations (75):
- United States (14):
  - University of California Irvine Medical Center, Irvine, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Wellstar MCG Augusta University, Augusta, Georgia
  - Northwestern University - Pulmonary and Critical Care Medicine, Chicago, Illinois
  - University of Louisville Hospital - Jewish Hospital, Louisville, Kentucky
  - University of Louisville-Jewish Hospital, Louisville, Kentucky
  - Mayo Clinic, Rochester, Minnesota
  - Hannibal Regional Hospital, Hannibal, Missouri
  - Bryan Medical Center, Lincoln, Nebraska
  - New York University Grossman School of Medicine, New York, New York
  - Penn State Health - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - McGovern Medical School - UT Physicians Pulmonary Medicine - Texas Medical Center, Houston, Texas
  - Baylor Scott & White Health, Temple, Texas
- Belgium (4):
  - HUB - Hôpital Erasme, Brussels
  - CHU Charleroi Marie Curie Hospital, Charleroi
  - Centre Hospitalier Regional de la Citadelle, Liège
  - Clinique Saint-Pierre Ottignies, Ottignies
- Bulgaria (3):
  - Acibadem City Clinic UMHAT Tokuda - Sofia, Sofia
  - Military Medical Academy, Sofia
  - UMHAT "Alexandrovska" EAD, Sofia
- Canada (11):
  - Foothills Medical Centre, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Grey Nuns Hospital, Edmonton, Alberta
  - Lions Gate Hospital, North Vancouver, British Columbia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network (UHN)-Toronto General Hospital (TGH), Toronto, Ontario
  - McGill University Health Centre - Royal Victoria Hospital (MUHC-RVH), Montreal, Quebec
  - Centre intégré universitaire de santé et services sociaux du nord de l'île de Montréal-Hôpital du Sacré de Montréal (CIUSSS-NÎM-HSCM), Montreal, Quebec
  - Peter Lougheed Centre, Calgary
  - Rocky View General Hospital, Calgary
  - South Health Campus, Calgary
- Czechia (3):
  - St. Anne's University Hospital, Brno
  - University Hospital Královské Vinohrady, Prague
  - General University Hospital, Prague
- France (8):
  - Centre Hospitalier Departemental (CHD) Vendee, La Roche-sur-Yon
  - Hôpital du Kremlin Bicêtre, APHP, Le Kremlin-Bicêtre
  - Centre Hospitalier de Melun-Senart, Melun
  - CHU Nantes, Nantes
  - Centre Hospitalier Lyon Sud, Oullins-Pierre-Bénite
  - Hopital Pitie-Salpetriere, Paris
  - Tenon Hospital, Paris
  - Nouvel Hopital Civil, Strasbourg
- Germany (3):
  - Saarland University Hospital, Homburg
  - Jena University Hospital, Jena
  - University Hospital LMU Munich, Munich
- Hungary (7):
  - National Institute of Pulmonology, Budapest
  - Petz Aladár University Teaching Hospital, Győr
  - Szent Damján Greek Catholic Hospital, Kisvárda
  - Szabolcs-Szatmar-Bereg County Teaching Hospital, Andras Josa Hospital, Nyíregyháza
  - Hospital of Siofok, Siófok
  - Teaching Hospital of Vas County, Szombathely
  - Ferenc Csolnoky Hospital of Veszprem County, Veszprém
- Italy (2):
  - Asst-Spedali Civili di Brescia, Brescia
  - Fondazione Policlinico A. Gemelli IRCCS, Rome
- Netherlands (5):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Gelre Hospitals, Department of ICU, Apeldoorn
  - Gelderse Vallei Hospital, Ede
  - Medisch Spectrum Twente, Enschede
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
- Romania (4):
  - University Hospital of Bucharest, Bucharest
  - Spital Universitar de Urgenta ELIAS (University Emergency Hospital Elias), Bucharest
  - County Clinical Hospital Tirgu Mures, Târgu Mureş
  - Clinical County Hospital Timisoara, Timișoara
- Spain (8):
  - Hospital Clínic Barcelona, Barcelona
  - University Hospital of Bucharest, Barcelona
  - Bellvitge University Hospital, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de Getafe, Madrid
  - Clínico San Carlos, Madrid
  - Hospital Universitari de Tarragona Joan XXIII, Tarragona
  - Hospital Universitari Sant Joan de Reus, Tarragona
- United Kingdom (3):
  - University Hospital of Wales, Cardiff
  - Derriford Hospital (University Hospitals Plymouth Hospital Trust), Plymouth
  - Pinderfields Hospital (Mid Yorkshire Teaching NHS Trust), Wakefield

IPD SHARING:
Plan to Share IPD: Yes